CLINICAL TRIAL: NCT02789111
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Alvimopan in Major Spine Surgery
Brief Title: Trial of Alvimopan in Major Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Bhiken I. Naik, MD, Anesthesiology attending, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18781
Record Dates: First submitted 2016-05-10; First posted 2016-06-02 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alvimopan (Active Comparator): 12 mg alvimopan twice a day (either by mouth or by (NG) nasogastric tube) for up to seven days post-operatively, or until the time of discharge, whichever occurs first, to a maximum of 15 doses.
  Interventions: Drug: Alvimopan
- Placebo (Placebo Comparator): Placebo twice a day (either by mouth or by (NG) nasogastric tube) for up to seven days post-operatively, or until the time of discharge, whichever occurs first, to a maximum of 15 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan — Alviimopan 12 mg twice daily up to 15 doses
  Other Names: Entereg
  Arms: Alvimopan
Drug: Placebo — Placebo twice daily up to 15 doses
  Arms: Placebo

SUMMARY:
The Investigator has chosen to study the reconstructive spinal surgery patient population because it is believed that the use of alvimopan in these patients at the University of Virginia will give the scientific community significant insight into the broader applicability of this drug into other surgical populations, the impact of this drug on the perception of pain (as opposed to simply the consumption of opioids), and its impact on total hospital charges, resource utilization, and functional outcomes.

DETAILED DESCRIPTION:
Pain control following major spine surgery is difficult to achieve. Opiates are often necessary in high doses, and may be associated with significant side effects. Such side effects may include urinary retention, altered mental status, depressed respiratory drive, and constipation, and may lead to reduced nutritional intake in the postoperative period. Importantly, post-operative nutrition may impact the incidence of complications following spine surgery.1 Alvimopan is a peripheral-acting opiate antagonist designed to decrease the gastrointestinal complications of perioperative systemic opioid administration.

Pain control following major spine surgery is difficult to achieve. Opiates are often necessary in high doses, and may be associated with significant side effects including constipation. Alvimopan is a drug approved by the Food and Drug Administration (FDA) and is used to help the bowel recover more quickly in patients who are having bowel surgery, so that they can eat solid foods and have regular bowel movements. Alvimopan is in a class of medications called peripherally acting mu-opioid receptor antagonists. It works by protecting the bowel from the constipation effects of opioid (narcotic) medications that are used to treat pain after surgery.

The purpose of this study is to determine if the use of alvimopan in major spine surgery reduces the time to first bowel movement. By assessing the use of alvimopan in reconstructive spinal surgery patients, researchers hope to give the scientific community insight into the broader use of this drug in other surgical populations, as well as gathering information on the impact of hospital charges and overall post-operative patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Major spine surgery scheduled as part of clinical care
* 18-80 years

Exclusion Criteria:

* More than three doses of any opioid within one week of surgery
* Pregnancy
* Prisoners
* Unable to provide consent
* Emergency surgery
* Chronic kidney disease stage 5 (GFR < 15 ml/min)
* Severe hepatic impairment
* Recent myocardial infarction (within the last 3 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhiken Naik, MBBCh, Principal Investigator — Anesthesiology Attending
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stambough JL, Beringer D. Postoperative wound infections complicating adult spine surgery. J Spinal Disord. 1992 Sep;5(3):277-85. doi: 10.1097/00002517-199209000-00005. PMID 1520986
- [Background] Crawford MW, Hickey C, Zaarour C, Howard A, Naser B. Development of acute opioid tolerance during infusion of remifentanil for pediatric scoliosis surgery. Anesth Analg. 2006 Jun;102(6):1662-7. doi: 10.1213/01.ane.0000216036.95705.c2. PMID 16717305
- [Background] Guignard B, Bossard AE, Coste C, Sessler DI, Lebrault C, Alfonsi P, Fletcher D, Chauvin M. Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology. 2000 Aug;93(2):409-17. doi: 10.1097/00000542-200008000-00019. PMID 10910490
- [Background] Rauf K, Vohra A, Fernandez-Jimenez P, O'Keeffe N, Forrest M. Remifentanil infusion in association with fentanyl-propofol anaesthesia in patients undergoing cardiac surgery: effects on morphine requirement and postoperative analgesia. Br J Anaesth. 2005 Nov;95(5):611-5. doi: 10.1093/bja/aei237. Epub 2005 Sep 9. PMID 16155034
- [Background] Cortinez LI, Brandes V, Munoz HR, Guerrero ME, Mur M. No clinical evidence of acute opioid tolerance after remifentanil-based anaesthesia. Br J Anaesth. 2001 Dec;87(6):866-9. doi: 10.1093/bja/87.6.866. PMID 11878688
- [Background] Fletcher D, Pinaud M, Scherpereel P, Clyti N, Chauvin M. The efficacy of intravenous 0.15 versus 0.25 mg/kg intraoperative morphine for immediate postoperative analgesia after remifentanil-based anesthesia for major surgery. Anesth Analg. 2000 Mar;90(3):666-71. doi: 10.1097/00000539-200003000-00029. PMID 10702454
- [Background] Lee LH, Irwin MG, Lui SK. Intraoperative remifentanil infusion does not increase postoperative opioid consumption compared with 70% nitrous oxide. Anesthesiology. 2005 Feb;102(2):398-402. doi: 10.1097/00000542-200502000-00024. PMID 15681957
- [Background] Bell TJ, Poston SA, Kraft MD, Senagore AJ, Delaney CP, Techner L. Economic analysis of alvimopan in North American Phase III efficacy trials. Am J Health Syst Pharm. 2009 Aug 1;66(15):1362-8. doi: 10.2146/ajhp080329. PMID 19635772
- [Background] Delaney CP, Weese JL, Hyman NH, Bauer J, Techner L, Gabriel K, Du W, Schmidt WK, Wallin BA; Alvimopan Postoperative Ileus Study Group. Phase III trial of alvimopan, a novel, peripherally acting, mu opioid antagonist, for postoperative ileus after major abdominal surgery. Dis Colon Rectum. 2005 Jun;48(6):1114-25; discussion 1125-6; author reply 1127-9. doi: 10.1007/s10350-005-0035-7. PMID 15906123
- [Background] Ludwig K, Enker WE, Delaney CP, Wolff BG, Du W, Fort JG, Cherubini M, Cucinotta J, Techner L. Gastrointestinal tract recovery in patients undergoing bowel resection: results of a randomized trial of alvimopan and placebo with a standardized accelerated postoperative care pathway. Arch Surg. 2008 Nov;143(11):1098-105. doi: 10.1001/archsurg.143.11.1098. PMID 19015469
- [Background] Viscusi ER, Goldstein S, Witkowski T, Andonakakis A, Jan R, Gabriel K, Du W, Techner L, Wallin B. Alvimopan, a peripherally acting mu-opioid receptor antagonist, compared with placebo in postoperative ileus after major abdominal surgery: results of a randomized, double-blind, controlled study. Surg Endosc. 2006 Jan;20(1):64-70. doi: 10.1007/s00464-005-0104-y. Epub 2005 Dec 7. PMID 16333556
- [Background] Wolff BG, Michelassi F, Gerkin TM, Techner L, Gabriel K, Du W, Wallin BA; Alvimopan Postoperative Ileus Study Group. Alvimopan, a novel, peripherally acting mu opioid antagonist: results of a multicenter, randomized, double-blind, placebo-controlled, phase III trial of major abdominal surgery and postoperative ileus. Ann Surg. 2004 Oct;240(4):728-34; discussion 734-5. doi: 10.1097/01.sla.0000141158.27977.66. PMID 15383800
- [Background] Herzog TJ, Coleman RL, Guerrieri JP Jr, Gabriel K, Du W, Techner L, Fort JG, Wallin B. A double-blind, randomized, placebo-controlled phase III study of the safety of alvimopan in patients who undergo simple total abdominal hysterectomy. Am J Obstet Gynecol. 2006 Aug;195(2):445-53. doi: 10.1016/j.ajog.2006.01.039. Epub 2006 Apr 19. PMID 16626607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-nine opioid-naive participants undergoing spine surgery between 2016 and 2018 with neurological monitoring were screened and included for eligibility. A total of 24 patients were assigned to the active group and 25 were assigned to the placebo group. One patient from the alvimopan group had surgery canceled, and thus was excluded from further analysis. In the placebo arm, 4 patients were recruited but withdrew from the study.
Pre-assignment Details: All 49 consented participants were assigned to an arm.
Period: Overall Study
Arm/Group | Alvimopan | Placebo
Started | 24 | 25
Completed | 23 | 21
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvimopan | Placebo | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Categorical [Count of Participants; unit: Participants] — Population: subjects who withdrew or did not have surgery were not analyzed
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 10 | 9 | 19
    >=65 years | 13 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants] — ONLY subjects that completed were analyzed Population: only subjects that completed were analyzed
  Participants
    Female | 14 | 9 | 23
    Male | 9 | 11 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to First Bowel Movement
Description: time to first bowel movement after surgery
Time Frame: Time to event( up to 7 days); From date of day of surgery until the date of first documented bowel movement
Measure: Mean (Full Range); unit: hours
Arm/Group | Alvimopan | Placebo
Number analyzed (Participants) | 23 | 20
hours | 50 [22 to 80] | 64 [40 to 114]

2. Secondary Outcome: Time to Resumption of PO Intake
Description: time to resumption oral intake after surgery
Time Frame: time to event ( up to 7 days); From date of day of surgery until the date of first documented PO intake
Population: Placebo vs. Alvimopan
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Placebo: Placebo group
- Alvimopan: Alvimopan group
Arm/Group | Placebo | Alvimopan
Number analyzed (Participants) | 20 | 23
hours | 17 [3 to 46] | 14.5 [3 to 25]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of surgery until 6 weeks after hospital discharge.
Arm/Group | Alvimopan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT02789111/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT02789111/ICF_001.pdf